CLINICAL TRIAL: NCT02074553
Title: A Randomized, Open-Label, Single Dose, Cross-Over Study to Investigate the Bioequivalence of Three RO5424802 Test Formulations Versus a Reference Formulation Following Oral Administration in Healthy Subjects
Brief Title: A Cross-over Study Examining the Bioequivalence of 3 Test Formulations to a Reference Formulation of Alectinib (RO5424802) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NP29040
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-03

CONDITIONS: Healthy Volunteer

ARMS (4):
- Ro542-4802/F03;Ro542-4802/F07;Ro542-4802/F14;Ro542-4802/F08 (Experimental): Participants will receive Ro542-4802/F03 (containing 50% SLS) capsules orally on Day 1 of first intervention period; then Ro542-4802/F07 (containing 25% SLS) capsules orally on Day 1 of second intervention period; then Ro542-4802/F14 (containing 12.5% SLS) capsules orally on Day 1 of third intervention period; followed by Ro542-4802/F08 (containing 3% SLS) capsules orally on Day 1 of fourth intervention period during both fasted (Part 1) and fed (Part 2) conditions. A washout period of at least 10 days will be maintained between each period.
  Interventions: Drug: Ro542-4802/F03 (Reference); Drug: Ro542-4802/F07 (Test); Drug: Ro542-4802/F08 (Test); Drug: Ro542-4802/F14 (Test)
- Ro542-4802/F07;Ro542-4802/F08;Ro542-4802/F03;Ro542-4802/F14 (Experimental): Participants will receive Ro542-4802/F07 (containing 25% SLS) capsules orally on Day 1 of first intervention period; then Ro542-4802/F08 (containing 3% SLS capsules orally on Day 1 in second intervention period; then Ro542-4802/F03 (containing 50% SLS) (containing 12.5% SLS) capsules orally on Day 1 of third intervention period; followed by Ro542-4802/F14 (containing 12.5% SLS) capsules orally on Day 1 of the fourth intervention period during both fasted (Part 1) and fed (Part 2) conditions. A washout period of at least 10 days will be maintained between each period.
  Interventions: Drug: Ro542-4802/F03 (Reference); Drug: Ro542-4802/F07 (Test); Drug: Ro542-4802/F08 (Test); Drug: Ro542-4802/F14 (Test)
- Ro542-4802/F08;Ro542-4802/F14;Ro542-4802/F07;Ro542-4802/F03 (Experimental): Participants will receive Ro542-4802/F08 (containing 3% SLS) capsules orally on Day 1 of first intervention period; then Ro542-4802/F14 (containing 12.5% SLS) capsules orally on Day 1 in second intervention period; then Ro542-4802/F07 (containing 25% SLS) capsules orally on Day 1 of third intervention period; followed by Ro542-4802/F03 (containing 50% SLS) capsules orally on Day 1 of the fourth intervention period during both fasted (Part 1) and fed (Part 2) conditions. A washout period of at least 10 days will be maintained between each period.
  Interventions: Drug: Ro542-4802/F03 (Reference); Drug: Ro542-4802/F07 (Test); Drug: Ro542-4802/F08 (Test); Drug: Ro542-4802/F14 (Test)
- Ro542-4802/F14;Ro542-4802/F03;Ro542-4802/F08;Ro542-4802/F07 (Experimental): Participants will receive Ro542-4802/F14 (containing 12.5% SLS) capsules orally on Day 1 of first intervention period; then Ro542-4802/F03 (containing 50% SLS) capsules orally on Day 1 in second intervention period; then Ro542-4802/F08 (containing 3% SLS) capsules orally on Day 1 of third intervention period; followed by Ro542-4802/F07 (containing 25% SLS) capsules orally on Day 1 of the fourth intervention period during both fasted (Part 1) and fed (Part 2) conditions. A washout period of at least 10 days will be maintained between each period.
  Interventions: Drug: Ro542-4802/F03 (Reference); Drug: Ro542-4802/F07 (Test); Drug: Ro542-4802/F08 (Test); Drug: Ro542-4802/F14 (Test)

INTERVENTIONS:
Drug: Ro542-4802/F03 (Reference) — Participants will receive Ro542-4802/F03 (containing 50% SLS) 600 mg capsules orally on Day 1.
Drug: Ro542-4802/F07 (Test) — Participants will receive Ro542-4802/F07 (containing 25% SLS) 600 mg capsules orally on Day 1.
Drug: Ro542-4802/F08 (Test) — Participants will receive Ro542-4802/F08 (containing 3% SLS) 600 mg capsules orally on Day 1.
Drug: Ro542-4802/F14 (Test) — Participants will receive Ro542-4802/F14 (containing 12.5% SLS) 600 mg capsules orally on Day 1.

SUMMARY:
This 2-part, single center, open-label, randomized, single-dose, 4-sequence, 4-period cross-over study will compare the bioequivalence of three test RO5424802 capsule formulations with the reference capsule formulation in healthy adult volunteers. All participants in both fasted (Part 1) and fed (Part 2) conditions of the study will receive each of 4 treatments (Ro542-4802/F03 [RO5424802 with 50 percentage (%) sodium lauryl sulfate (SLS) (reference)], Ro542-4802/F07 [RO5424802 with 25% SLS (test)], Ro542-4802/F14 [RO5424802 with 12.5% SLS (test)] and Ro542-4802/F08 [RO5424802 with 3% SLS (test)] in a randomized sequence. Each treatment will be given as a single 600 milligrams (mg) oral administration in an upright position on Day 1 after an overnight fast, followed by a 10-day washout period. Total time on study is expected to last up to 75 days, for each enrolled participant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and surgically sterile or post-menopausal female participants 18-55 years of age
* Body mass index (BMI) between 18 to 32 kilograms per meter-squared (kg/m^2)
* Non-smoking participants and former smoking participants (who have not smoked for the past six months before first dosing)
* Male participants and their partners of child-bearing potential must be willing to use two effective contraceptive methods as defined by protocol
* Willing to abstain from xanthine-containing beverages and food (coffee, tea, cola, chocolate, and "energy drinks") from 72 hours prior to Day -1 through the study
* Willing to abstain from grapefruit, pomelo, star fruit or Seville orange containing products from day 7 prior study start until study end
* Willing to avoid prolonged sun exposure while taking RO5424802 and through follow-up

Exclusion Criteria:

* Pregnant or lactating women, men with female partners who are pregnant or lactating, or women of child bearing potential
* Clinically significant abnormalities on physical examination, vital signs, or laboratory test results during screening or prior to admission to the study unit
* Positive test for drugs of abuse, alcohol or cotinine test at screening or prior to admission to the study unit or suspicion of regular consumption of drug(s) of abuse
* History of recent alcohol consumption exceeding 2 standard drinks per day on average. Alcohol consuming is prohibited from 72 hours prior to study start until the end of the study
* Participants with any risk factors or family history for QT/QTcF and electrocardiogram (ECG) abnormalities
* A history of any concurrent clinically significant hematologic, renal, hepatic, pulmonary, neurological, psychiatric, allergies, gastrointestinal, metabolic or endocrine disorder, or cardiovascular disease or infections
* Positive screening test for hepatitis B, C, or human immunodeficiency virus (HIV)
* Use of any medications (prescriptions or over-the-counter), within 2 weeks or 5 half-lives (whichever is longer) before the first dose of study medication with exception of acetaminophen up to 2 grams (g) per day up to 48 hours prior to dosing, not to exceed 4 g total during the week prior to dosing
* Routine or chronic use of more than 2 g of acetaminophen daily
* Use of any herbal supplements (for example, St. John's Wort) or any metabolic inducers within 4 weeks or 5 half-lives (whichever is longer) before the first dose of study medication, including but not limited to the following drugs: rifampin, rifabutin, glucocorticoids, carbamazepine, phenytoin, and phenobarbital
* Strenuous activity, sunbathing or contact sports are not allowed from 4 days prior to study start until the end of the study
* Participation in an investigational drug or device study within 45 days or 5 half-lives (whichever time period is longer), or 6 months for biologic therapies, prior to first dosing
* Donation of blood over 450 milliliters (mL) within 45 days prior to screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1 (Fasted): Treatment A Then B Then C Then D: Participants following an overnight fast of at least 10 hours received 600 milligram (mg) of alectinib (RO5424802) as a capsule formulation (four 150 mg capsules) orally in Part 1 of the study according to following treatment sequences. Treatment A (Reference Treatment: formulation containing 50 percent [%]sodium lauryl sulfate [SLS]) on Day 1 of the first intervention period; then Treatment B (Test Treatment: formulation containing 25% SLS) on Day 1 of second intervention period (Day 11); then Treatment C (Test Treatment: formulation containing 12.5% SLS) on Day 1 of third intervention period (Day 21); followed by Treatment D (Test Treatment: formulation containing 3% SLS) on Day 1 of fourth intervention period (Day 31). A washout period of at least 10 days was maintained between each intervention period.
- Part 1 (Fasted): Treatment B Then D Then A Then C: Participants following an overnight fast of at least 10 hours received 600 mg of alectinib as a capsule formulation orally in Part 1 of the study according to following treatment sequences. Treatment B (formulation containing 25% SLS) on Day 1 of the first intervention period; then Treatment D (formulation containing 3% SLS) on Day 1 of second intervention period (Day 11); then Treatment A (formulation containing 50% SLS) on Day 1 of third intervention period (Day 21); followed by Treatment C (formulation containing 12.5% SLS) on Day 1 of fourth intervention period (Day 31). A washout period of at least 10 days was maintained between each intervention period.
- Part 1 (Fasted): Treatment C Then A Then D Then B: Participants following an overnight fast of at least 10 hours received 600 mg of alectinib as a capsule formulation orally in Part 1 of the study according to following treatment sequences. Treatment C (formulation containing 12.5% SLS) on Day 1 of the first intervention period; then Treatment A (formulation containing 50% SLS) on Day 1 of second intervention period (Day 11); then Treatment D (formulation containing 3% SLS) on Day 1 of third intervention period (Day 21); followed by Treatment B (formulation containing 25% SLS) on Day 1 of fourth intervention period (Day 31). A washout period of at least 10 days was maintained between each intervention period.
- Part 1 (Fasted): Treatment D Then C Then B Then A: Participants following an overnight fast of at least 10 hours received 600 mg of alectinib as a capsule formulation orally in Part 1 of the study according to following treatment sequences. Treatment D (formulation containing 3% SLS) on Day 1 of the first intervention period; then Treatment C (formulation containing 12.5% SLS) on Day 1 of second intervention period (Day 11); then Treatment B (formulation containing 25% SLS) on Day 1 of third intervention period (Day 21); followed by Treatment A (formulation containing 50% SLS) on Day 1 of fourth intervention period (Day 31). A washout period of at least 10 days was maintained between each intervention period.
- Part 2 (Fed): Treatment A Then B Then C Then D: Participants following an overnight fast of at least 10 hours ate a high-fat, high-calorie meal in 30 minutes or less and 30 minutes after start of the meal received 600 mg of alectinib as a capsule formulation orally in Part 2 of the study according to following treatment sequences. Treatment A (formulation containing 50% SLS) on Day 1 of the first intervention period; then Treatment B (formulation containing 25% SLS) on Day 1 of second intervention period (Day 11); then Treatment C (formulation containing 12.5% SLS) on Day 1 of third intervention period (Day 21); followed by Treatment D (formulation containing 3% SLS) on Day 1 of fourth intervention period (Day 31). A washout period of at least 10 days was maintained between each intervention period.
- Part 2 (Fed): Treatment B Then D Then A Then C: Participants following an overnight fast of at least 10 hours ate a high-fat, high-calorie meal in 30 minutes or less and 30 minutes after start of the meal received 600 mg of alectinib as a capsule formulation orally in Part 2 of the study according to following treatment sequences. Treatment B (formulation containing 25% SLS) on Day 1 of the first intervention period; then Treatment D (formulation containing 3% SLS) on Day 1 of second intervention period (Day 11); then Treatment A (formulation containing 50% SLS) on Day 1 of third intervention period (Day 21); followed by Treatment C (formulation containing 12.5% SLS) on Day 1 of fourth intervention period (Day 31). A washout period of at least 10 days was maintained between each intervention period.
- Part 2 (Fed): Treatment C Then A Then D Then B: Participants following an overnight fast of at least 10 hours ate a high-fat, high-calorie meal in 30 minutes or less and 30 minutes after start of the meal received 600 mg of alectinib as a capsule formulation orally in Part 2 of the study according to following treatment sequences. Treatment C (formulation containing 12.5% SLS) on Day 1 of the first intervention period; then Treatment A (formulation containing 50% SLS) on Day 1 of second intervention period (Day 11); then Treatment D (formulation containing 3% SLS) on Day 1 of third intervention period (Day 21); followed by Treatment B (formulation containing 25% SLS) on Day 1 of fourth intervention period (Day 31). A washout period of at least 10 days was maintained between each intervention period.
- Part 2 (Fed): Treatment D Then C Then B Then A: Participants following an overnight fast of at least 10 hours ate a high-fat, high-calorie meal in 30 minutes or less and 30 minutes after start of the meal received 600 mg of alectinib as a capsule formulation orally in Part 2 of the study according to following treatment sequences. Treatment D (formulation containing 3% SLS) on Day 1 of the first intervention period; then Treatment C (formulation containing 12.5% SLS) on Day 1 of second intervention period (Day 11); then Treatment B (formulation containing 25% SLS) on Day 1 of third intervention period (Day 21); followed by Treatment A (formulation containing 50% SLS) on Day 1 of fourth intervention period (Day 31). A washout period of at least 10 days was maintained between each intervention period.
Period: Intervention Period 1
Arm/Group | Part 1 (Fasted): Treatment A Then B Then C Then D | Part 1 (Fasted): Treatment B Then D Then A Then C | Part 1 (Fasted): Treatment C Then A Then D Then B | Part 1 (Fasted): Treatment D Then C Then B Then A | Part 2 (Fed): Treatment A Then B Then C Then D | Part 2 (Fed): Treatment B Then D Then A Then C | Part 2 (Fed): Treatment C Then A Then D Then B | Part 2 (Fed): Treatment D Then C Then B Then A
Started | 12 | 12 | 12 | 13 | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Family Emergency | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | Part 1 (Fasted): Treatment A Then B Then C Then D | Part 1 (Fasted): Treatment B Then D Then A Then C | Part 1 (Fasted): Treatment C Then A Then D Then B | Part 1 (Fasted): Treatment D Then C Then B Then A | Part 2 (Fed): Treatment A Then B Then C Then D | Part 2 (Fed): Treatment B Then D Then A Then C | Part 2 (Fed): Treatment C Then A Then D Then B | Part 2 (Fed): Treatment D Then C Then B Then A
Started | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Completed | 11 | 12 | 12 | 11 | 12 | 11 | 12 | 12
Not Completed | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Intervention Period 2
Arm/Group | Part 1 (Fasted): Treatment A Then B Then C Then D | Part 1 (Fasted): Treatment B Then D Then A Then C | Part 1 (Fasted): Treatment C Then A Then D Then B | Part 1 (Fasted): Treatment D Then C Then B Then A | Part 2 (Fed): Treatment A Then B Then C Then D | Part 2 (Fed): Treatment B Then D Then A Then C | Part 2 (Fed): Treatment C Then A Then D Then B | Part 2 (Fed): Treatment D Then C Then B Then A
Started | 11 | 12 | 12 | 11 | 12 | 11 | 12 | 12
Completed | 11 | 12 | 12 | 11 | 12 | 11 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Part 1 (Fasted): Treatment A Then B Then C Then D | Part 1 (Fasted): Treatment B Then D Then A Then C | Part 1 (Fasted): Treatment C Then A Then D Then B | Part 1 (Fasted): Treatment D Then C Then B Then A | Part 2 (Fed): Treatment A Then B Then C Then D | Part 2 (Fed): Treatment B Then D Then A Then C | Part 2 (Fed): Treatment C Then A Then D Then B | Part 2 (Fed): Treatment D Then C Then B Then A
Started | 11 | 12 | 12 | 11 | 12 | 11 | 12 | 12
Completed | 11 | 12 | 11 | 11 | 12 | 10 | 11 | 12
Not Completed | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 3
Arm/Group | Part 1 (Fasted): Treatment A Then B Then C Then D | Part 1 (Fasted): Treatment B Then D Then A Then C | Part 1 (Fasted): Treatment C Then A Then D Then B | Part 1 (Fasted): Treatment D Then C Then B Then A | Part 2 (Fed): Treatment A Then B Then C Then D | Part 2 (Fed): Treatment B Then D Then A Then C | Part 2 (Fed): Treatment C Then A Then D Then B | Part 2 (Fed): Treatment D Then C Then B Then A
Started | 11 | 12 | 11 | 11 | 12 | 10 | 11 | 12
Completed | 11 | 12 | 11 | 11 | 12 | 10 | 11 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3
Arm/Group | Part 1 (Fasted): Treatment A Then B Then C Then D | Part 1 (Fasted): Treatment B Then D Then A Then C | Part 1 (Fasted): Treatment C Then A Then D Then B | Part 1 (Fasted): Treatment D Then C Then B Then A | Part 2 (Fed): Treatment A Then B Then C Then D | Part 2 (Fed): Treatment B Then D Then A Then C | Part 2 (Fed): Treatment C Then A Then D Then B | Part 2 (Fed): Treatment D Then C Then B Then A
Started | 11 | 12 | 11 | 11 | 12 | 10 | 11 | 12
Completed | 11 | 12 | 11 | 11 | 12 | 10 | 11 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Intervention Period 4
Arm/Group | Part 1 (Fasted): Treatment A Then B Then C Then D | Part 1 (Fasted): Treatment B Then D Then A Then C | Part 1 (Fasted): Treatment C Then A Then D Then B | Part 1 (Fasted): Treatment D Then C Then B Then A | Part 2 (Fed): Treatment A Then B Then C Then D | Part 2 (Fed): Treatment B Then D Then A Then C | Part 2 (Fed): Treatment C Then A Then D Then B | Part 2 (Fed): Treatment D Then C Then B Then A
Started | 11 | 12 | 11 | 11 | 12 | 10 | 11 | 11
Completed | 11 | 12 | 11 | 11 | 12 | 10 | 11 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of the study drug and had at least 1 safety assessment after dosing.
Groups:
- Part 1 (Fasted): Study Population: Participants following an overnight fast of at least 10 hours received alectinib 600 mg capsules orally as Treatment A, B, C, and D according to any of the four treatment sequences in Part 1 of the study.
- Part 2 (Fed): Study Population: Participants following an overnight fast of at least 10 hours ate the high-fat, high-calorie meal in 30 minutes or less and 30 minutes after the start of the meal received alectinib 600 mg capsules orally as Treatment A, B, C, and D according to any of the four treatment sequences in Part 2 of the study.
- Total: Total of all reporting groups
Arm/Group | Part 1 (Fasted): Study Population | Part 2 (Fed): Study Population | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (10.01) | 36.1 (10.49) | 36.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 41 | 42 | 83

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Extrapolated Infinite Time (AUC[0-inf]) of Alectinib
Description: AUC(0-inf) is the area under the alectinib plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). AUC is a measure of the plasma concentration of a drug over time. AUC(0-inf) is presented in nanogram times (*) hour per milliliter (ng*hour/mL).
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: The Pharmacokinetic (PK) analysis set included all participants who received the reference formulation 50% SLS alectinib (Treatment A) and at least 1 test formulation (Treatments B, C, or D) and provided adequate PK assessments.
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Groups:
- Part 1 (Fasted): Treatment A: Participants following an overnight fast of at least 10 hours received alectinib 600 mg capsules orally as Treatment A (formulation containing 50% SLS) on Day 1 of any of the four intervention periods in Part 1.
- Part 1 (Fasted): Treatment B: Participants following an overnight fast of at least 10 hours received alectinib 600 mg capsules orally as Treatment B (formulation containing 25% SLS) on Day 1 of any of the four intervention periods in Part 1.
- Part 1 (Fasted): Treatment C: Participants following an overnight fast of at least 10 hours received alectinib 600 mg capsules orally as Treatment C (formulation containing 12.5% SLS) on Day 1 of any of the four intervention periods in Part 1.
- Part 1 (Fasted): Treatment D: Participants following an overnight fast of at least 10 hours received alectinib 600 mg capsules orally as Treatment D (formulation containing 3% SLS) on Day 1 of any of the four intervention periods in Part 1.
- Part 2 (Fed): Treatment A: Participants following an overnight fast of at least 10 hours ate the high-fat, high-calorie meal in 30 minutes or less and 30 minutes after the start of the meal received alectinib 600 mg capsules orally as Treatment A (formulation containing 50% SLS) on Day 1 of any of the four intervention periods in Part 2.
- Part 2 (Fed): Treatment B: Participants following an overnight fast of at least 10 hours ate the high-fat, high-calorie meal in 30 minutes or less and 30 minutes after the start of the meal received alectinib 600 mg capsules orally as Treatment B (formulation containing 25% SLS) on Day 1 of any of the four intervention periods in Part 2.
- Part 2 (Fed): Treatment C: Participants following an overnight fast of at least 10 hours ate the high-fat, high-calorie meal in 30 minutes or less and 30 minutes after the start of the meal received alectinib 600 mg capsules orally as Treatment C (formulation containing 12.5% SLS) on Day 1 of any of the four intervention periods in Part 2.
- Part 2 (Fed): Treatment D: Participants following an overnight fast of at least 10 hours ate the high-fat, high-calorie meal in 30 minutes or less and 30 minutes after the start of the meal received alectinib 600 mg capsules orally as Treatment D (formulation containing 3% SLS) on Day 1 of any of the four intervention periods in Part 2.
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
ng*hour/mL | 1920 (1000) | 1840 (754) | 1850 (841) | 1630 (792) | 5720 (1530) | 5050 (1200) | 4600 (1260) | 4580 (1240)
Statistical Analysis 1: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment B; Analysis of variance (ANOVA) (fixed factors: treatment, period, and treatment sequence; and random factor: participant) was applied to the log-transformed PK parameter, and then back transformed to provide geometric least square mean ratio (Test/Reference) and 90% confidence interval (CI); Test type: Non-Inferiority or Equivalence — Bioequivalence of the test formulation was concluded if its 90% CI was included in the bioequivalence range of 80% to 125%; Geometric Least Square Mean Ratio = 100.5, 90% CI 2-sided [93.14 to 108.44] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 2: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment C; ANOVA (fixed factors: treatment, period, and treatment sequence; and random factor: participant) was applied to the log-transformed PK parameter, and then back transformed to provide geometric least square mean ratio (Test/Reference) and 90% CI; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 97.82, 90% CI 2-sided [90.71 to 105.48] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 3: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 86.66, 90% CI 2-sided [80.32 to 93.5] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 4: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment B; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 88.62, 90% CI 2-sided [85.15 to 92.24] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 5: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 80.17, 90% CI 2-sided [77.08 to 83.39] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 6: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 79.95, 90% CI 2-sided [76.84 to 83.19] — The reported values are percentages of geometric least square mean ratio

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC[0-last]) of Alectinib
Description: AUC(0-last) is the area under the alectinib plasma concentration versus time curve from time zero to the time of last measured concentration of alectinib. AUC is a measure of the plasma concentration of a drug over time. AUC(0-last) is presented in ng*hour/mL.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
ng*hour/mL | 1790 (925) | 1680 (620) | 1620 (637) | 1380 (573) | 5540 (1460) | 4820 (1130) | 4370 (1170) | 4360 (1160)
Statistical Analysis 1: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment B; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 99.12, 90% CI 2-sided [91.83 to 106.99] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 2: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 93.79, 90% CI 2-sided [86.94 to 101.17] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 3: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 80.32, 90% CI 2-sided [74.41 to 86.7] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 4: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment B; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 87.42, 90% CI 2-sided [83.92 to 91.07] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 5: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 78.87, 90% CI 2-sided [75.76 to 82.11] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 6: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 78.66, 90% CI 2-sided [75.53 to 81.92] — The reported values are percentages of geometric least square mean ratio

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Alectinib
Description: Cmax is the maximum observed plasma alectinib concentration, presented in nanogram per milliliter (ng/mL).
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
ng/mL | 106 (53.3) | 91.7 (34.5) | 67.0 (23.6) | 42.2 (19.2) | 271 (81.8) | 232 (59.3) | 206 (50.4) | 204 (57.1)
Statistical Analysis 1: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment B; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 90.34, 90% CI 2-sided [82.33 to 99.12] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 2: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 66.28, 90% CI 2-sided [60.45 to 72.68] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 3: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 41.04, 90% CI 2-sided [37.40 to 45.03] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 4: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment B; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 86.30, 90% CI 2-sided [81.77 to 91.09] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 5: Comparison: Part 2 (Fed): Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 77.00, 90% CI 2-sided [73.01 to 81.20] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 6: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 75.65, 90% CI 2-sided [71.71 to 79.82] — The reported values are percentages of geometric least square mean ratio

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Alectinib
Description: Tmax is the time from alectinib administration to reach Cmax for alectinib.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
hours | 3.25 [1.50 to 12.0] | 3.00 [1.00 to 5.00] | 3.00 [2.00 to 6.00] | 4.00 [2.50 to 10.0] | 8.00 [4.05 to 18.0] | 8.00 [5.00 to 18.0] | 6.00 [4.00 to 12.0] | 6.00 [4.00 to 10.0]

5. Secondary Outcome: Cmax of RO5468924
Description: Cmax is the maximum observed plasma RO5468924 concentration, presented in ng/mL. RO5468924 is the major pharmacologically active metabolite of alectinib.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
ng/mL | 33.0 (15.4) | 30.7 (14.9) | 21.9 (8.94) | 11.3 (5.71) | 98.8 (28.6) | 92.2 (28.7) | 71.4 (20.6) | 65.2 (16.8)
Statistical Analysis 1: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment B; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 91.67, 90% CI 2-sided [82.34 to 102.05] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 2: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 67.24, 90% CI 2-sided [60.44 to 74.79] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 3: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 34.32, 90% CI 2-sided [30.83 to 38.21] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 4: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment B; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 95.15, 90% CI 2-sided [89.10 to 101.62] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 5: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 73.26, 90% CI 2-sided [68.67 to 78.16] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 6: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 67.76, 90% CI 2-sided [63.48 to 72.33] — The reported values are percentages of geometric least square mean ratio

6. Secondary Outcome: Tmax of RO5468924
Description: Tmax is the time from alectinib administration to reach Cmax for RO5468924 (the major pharmacologically active metabolite of alectinib).
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
hours | 8.00 [8.00 to 12.0] | 8.02 [6.00 to 12.1] | 8.00 [6.00 to 12.0] | 8.07 [4.00 to 12.1] | 12.0 [6.00 to 24.0] | 10.0 [5.03 to 24.0] | 8.02 [6.00 to 12.1] | 9.00 [5.00 to 24.0]

7. Secondary Outcome: AUC(0-inf) of RO5468924
Description: AUC(0-inf) is the area under the RO5468924 plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). RO5468924 is the major pharmacologically active metabolite of alectinib. AUC is a measure of the plasma concentration of a drug over time. AUC(0-inf) is presented in ng*hour/mL.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
ng*hour/mL | 968 (397) | 936 (419) | 754 (298) | 534 (279) | 3010 (819) | 2660 (687) | 2200 (578) | 2100 (543)
Statistical Analysis 1: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment B; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 95.77, 90% CI 2-sided [87.54 to 104.79] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 2: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 78.69, 90% CI 2-sided [71.97 to 86.04] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 3: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 53.91, 90% CI 2-sided [49.27 to 58.98] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 4: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment B; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 90.16, 90% CI 2-sided [86.14 to 94.37] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 5: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 73.76, 90% CI 2-sided [70.52 to 77.15] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 6: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 70.94, 90% CI 2-sided [67.80 to 74.22] — The reported values are percentages of geometric least square mean ratio

8. Secondary Outcome: AUC(0-last) of RO5468924
Description: AUC(0-last) is the area under the RO5468924 plasma concentration versus time curve from time zero to the time of last measured concentration of RO5468924. RO5468924 is the major pharmacologically active metabolite of alectinib. AUC is a measure of the plasma concentration of a drug over time. AUC(0-last) is presented in ng*hour/mL.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
ng*hour/mL | 876 (375) | 826 (376) | 641 (248) | 392 (199) | 2780 (773) | 2460 (669) | 2000 (531) | 1890 (477)
Statistical Analysis 1: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment B; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 93.05, 90% CI 2-sided [84.24 to 102.78] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 2: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 74.35, 90% CI 2-sided [67.37 to 82.06] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 3: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 43.94, 90% CI 2-sided [39.78 to 48.53] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 4: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment B; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 90.21, 90% CI 2-sided [86.12 to 94.49] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 5: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 72.72, 90% CI 2-sided [69.48 to 76.12] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 6: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 69.34, 90% CI 2-sided [66.23 to 72.61] — The reported values are percentages of geometric least square mean ratio

9. Secondary Outcome: Plasma Terminal Half-Life (t1/2) of Alectinib and RO5468924
Description: Plasma terminal half-life is the time measured during drug elimination phase for the plasma drug concentration to decrease by one half. RO5468924 is the major pharmacologically active metabolite of alectinib.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
hours
  Alectinib | 23.6 (11.1) | 24.3 (11.1) | 25.6 (11.2) | 28.8 (17.4) | 19.8 (6.56) | 21.3 (10.6) | 21.4 (10.3) | 21.9 (12.0)
  RO5468924 | 28.1 (8.29) | 30.7 (9.63) | 31.8 (12.7) | 41.7 (19.8) | 28.3 (6.79) | 27.4 (5.27) | 29.1 (7.13) | 31.0 (7.74)

10. Secondary Outcome: Elimination Rate Constant (Kel) of Alectinib and RO5468924
Description: First-order terminal elimination rate constant (Kel) was calculated as the negative slope of the linear regression of the terminal phase in plasma alectinib and RO5468924 concentration versus time profile using appropriate time points. RO5468924 is the major pharmacologically active metabolite of alectinib.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
1/hour
  Alectinib | 0.0340 (0.0113) | 0.0333 (0.0119) | 0.0312 (0.0108) | 0.0303 (0.0123) | 0.0371 (0.00732) | 0.0369 (0.0117) | 0.0371 (0.0117) | 0.0367 (0.0110)
  RO5468924 | 0.0267 (0.00750) | 0.0248 (0.00767) | 0.0240 (0.00654) | 0.0199 (0.00753) | 0.0256 (0.00493) | 0.0263 (0.00540) | 0.0252 (0.00618) | 0.0236 (0.00538)

11. Secondary Outcome: Total Molar Concentration of Alectinib and RO5468924 as Derived by AUC(0-inf)
Description: AUC(0-inf) is the area under the alectinib + RO5468924 (major pharmacologically active metabolite of alectinib) molar plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (0-inf). AUC is a measure of the plasma concentration of the alectinib + RO5468924 over time. AUC(0-inf) is presented in nanomoles times (*) hour per liter (nmol*hour/L).
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: nmol*hour/L
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
nmol*hour/L | 6040 (2870) | 5780 (2290) | 5450 (2310) | 4470 (2370) | 18400 (4600) | 16200 (3650) | 14300 (3570) | 14100 (3490)
Statistical Analysis 1: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment B; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 98.79, 90% CI 2-sided [91.25 to 106.95] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 2: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 91.58, 90% CI 2-sided [84.65 to 99.08] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 3: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 73.41, 90% CI 2-sided [67.81 to 79.47] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 4: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment B; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 88.81, 90% CI 2-sided [85.62 to 92.13] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 5: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 77.74, 90% CI 2-sided [74.99 to 80.60] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 6: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 76.65, 90% CI 2-sided [73.92 to 79.49] — The reported values are percentages of geometric least square mean ratio

12. Secondary Outcome: Total Molar Concentration of Alectinib and RO5468924 as Derived by Cmax
Description: Cmax is the maximum observed molar plasma concentration for alectinib + RO5468924 (major pharmacologically active metabolite of alectinib). Cmax is presented in nanomoles per liter (nmol/L).
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
nmol/L | 257 (123) | 221 (79.6) | 164 (52.6) | 106 (48.6) | 754 (209) | 662 (162) | 566 (138) | 548 (141)
Statistical Analysis 1: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment B; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 89.41, 90% CI 2-sided [81.7 to 97.84] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 2: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 66.84, 90% CI 2-sided [61.12 to 73.1] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 3: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 42.32, 90% CI 2-sided [38.68 to 46.32] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 4: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment B; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 88.76, 90% CI 2-sided [84.21 to 93.56] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 5: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 75.82, 90% CI 2-sided [71.99 to 79.86] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 6: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 73.26, 90% CI 2-sided [69.53 to 77.19] — The reported values are percentages of geometric least square mean ratio

13. Secondary Outcome: Total Molar Concentration of Alectinib and RO5468924 as Derived by AUC(0-last)
Description: AUC(0-last) is the area under the alectinib + RO5468924 (major pharmacologically active metabolite of alectinib) molar plasma concentration versus time curve from time zero to the time of last measured concentration of alectinib + RO5468924. AUC(0-last) is presented in nmol*hour/L.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: nmol*hour/L
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
nmol*hour/L | 5660 (2620) | 5310 (1980) | 4780 (1710) | 3740 (1560) | 17600 (4370) | 15400 (3500) | 13400 (3260) | 13200 (3200)
Statistical Analysis 1: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment B; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 97.23, 90% CI 2-sided [89.85 to 105.21] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 2: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 87.16, 90% CI 2-sided [80.59 to 94.26] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 3: Comparison: Part 1 (Fasted): Treatment A vs Part 1 (Fasted): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 67.86, 90% CI 2-sided [62.71 to 73.43] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 4: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment B; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 88.28, 90% CI 2-sided [85.06 to 91.63] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 5: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment C; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 76.79, 90% CI 2-sided [74.03 to 79.65] — The reported values are percentages of geometric least square mean ratio
Statistical Analysis 6: Comparison: Part 2 (Fed): Treatment A vs Part 2 (Fed): Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 75.43, 90% CI 2-sided [72.70 to 78.27] — The reported values are percentages of geometric least square mean ratio

14. Secondary Outcome: Apparent Oral Clearance (CL/F) of Alectinib
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: liters/hour
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
liters/hour | 377 (149) | 380 (152) | 383 (151) | 449 (199) | 113 (30.9) | 126 (31.5) | 141 (39.3) | 141 (40.2)

15. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Alectinib
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction of drug absorbed.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
liters | 12200 (6240) | 12200 (5120) | 12900 (4430) | 16500 (7300) | 3180 (1260) | 3730 (1530) | 4180 (1920) | 4290 (2240)

16. Secondary Outcome: Percent Extrapolated AUC(0-inf) (AUC%Extrap[0-inf]) for Alectinib and RO5468924
Description: The AUC%extrap(0-inf), that is, area obtained after extrapolation (extrap) from time to last quantifiable plasma concentration (Tlast) to infinity is calculated by using the formula AUC%extrap(0-inf) = 100*(AUC[0-inf] minus AUC[0-last])/AUC(0-inf); where AUC(0-inf) = Area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time and AUC(0-last) is area under the plasma concentration time-curve from zero (pre-dose) to the time of last measured concentration. The function of this parameter is to provide information about what percentage of the theoretical curve AUC(0-inf) was possible to determine experimentally (AUC0-last).
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: percent AUC
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
percent AUC
  Alectinib | 6.43 (4.06) | 7.45 (6.25) | 9.91 (8.08) | 12.5 (10.9) | 3.04 (2.57) | 4.24 (5.01) | 4.49 (4.86) | 4.52 (5.54)
  RO5468924 | 10.2 (3.67) | 12.6 (6.14) | 14.9 (6.89) | 26.0 (11.2) | 7.84 (2.57) | 7.84 (2.52) | 9.12 (3.39) | 9.94 (3.93)

17. Secondary Outcome: Adjusted r^2 Value (Rsq) for Regression Estimation of Kel for Alectinib and RO5468924
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: no units
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
no units
  Alectinib | 0.987 (0.0252) | 0.983 (0.0277) | 0.973 (0.0622) | 0.976 (0.0337) | 0.994 (0.00812) | 0.991 (0.0189) | 0.990 (0.0206) | 0.991 (0.0153)
  RO5468924 | 0.977 (0.0233) | 0.970 (0.0293) | 0.963 (0.0591) | 0.958 (0.0687) | 0.986 (0.0124) | 0.980 (0.0186) | 0.977 (0.0178) | 0.982 (0.0195)

18. Secondary Outcome: Molecular Weight Adjusted Metabolite to Parent (M/P) Ratio for AUC(0-inf)
Description: AUC(0-inf) is the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). AUC is a measure of the plasma concentration of the alectinib and RO5468924 (major pharmacologically active metabolite of alectinib) over time. The molecular weight adjusted M/P ratio (RO5468924/alectinib) for AUC(0-inf) is presented.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
ratio | 0.54 (0.0705) | 0.52 (0.0720) | 0.43 (0.0512) | 0.34 (0.0233) | 0.55 (0.0468) | 0.56 (0.0393) | 0.51 (0.0290) | 0.49 (0.0300)

19. Secondary Outcome: Molecular Weight Adjusted M/P Ratio for AUC(0-last)
Description: AUC(0-last) is the area under the plasma concentration versus time curve from time zero to the time of last measured concentration. AUC is a measure of the plasma concentration of the alectinib and RO5468924 (major pharmacologically active metabolite of alectinib) over time. The molecular weight adjusted M/P ratio (RO5468924/alectinib) for AUC(0-last) is presented.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
ratio | 0.52 (0.0708) | 0.49 (0.0838) | 0.41 (0.0458) | 0.29 (0.0347) | 0.52 (0.0474) | 0.54 (0.0384) | 0.48 (0.0264) | 0.46 (0.0237)

20. Secondary Outcome: Molecular Weight Adjusted M/P Ratio for Cmax
Description: Cmax is the maximum observed plasma concentration of the alectinib and RO5468924 (major pharmacologically active metabolite of alectinib). The molecular weight adjusted M/P ratio (RO5468924/alectinib) for Cmax is presented.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
ratio | 0.33 (0.0376) | 0.34 (0.0446) | 0.33 (0.0438) | 0.28 (0.0206) | 0.38 (0.0445) | 0.42 (0.0304) | 0.36 (0.0223) | 0.34 (0.0207)

21. Secondary Outcome: Time to Reach Last Quantifiable Plasma Concentration (Tlast) of Alectinib and RO5468924
Description: Tlast is the time from alectinib administration to reach last quantifiable concentration of alectinib and its major pharmacologically active metabolite RO5468924.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 60, 72, and 96 hours postdose
Population: PK analysis set
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 43 | 45 | 44
hours
  Alectinib | 96.0 [60.0 to 96.1] | 96.0 [60.0 to 96.1] | 96.0 [60.0 to 96.2] | 96.0 [60.0 to 96.1] | 96.0 [72.1 to 96.1] | 96.0 [72.0 to 96.1] | 96.0 [72.0 to 96.1] | 96.0 [72.0 to 96.2]
  RO5468924 | 96.0 [48.0 to 96.1] | 96.0 [48.0 to 96.0] | 96.0 [60.0 to 96.2] | 72.0 [36.0 to 96.2] | 96.0 [96.0 to 96.1] | 96.0 [96.0 to 96.1] | 96.0 [96.0 to 96.1] | 96.0 [96.0 to 96.2]

ADVERSE EVENTS:
Time Frame: Day 1 through follow-up (up to 47 days)
Description: Safety analysis set. An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A treatment-emergent AE (TEAE) was defined as an AE that began or worsened in severity on or after the first dose of the study drug.
Arm/Group | Part 1 (Fasted): Treatment A | Part 1 (Fasted): Treatment B | Part 1 (Fasted): Treatment C | Part 1 (Fasted): Treatment D | Part 2 (Fed): Treatment A | Part 2 (Fed): Treatment B | Part 2 (Fed): Treatment C | Part 2 (Fed): Treatment D
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/45 | 0/46 | 0/47 | 0/45 | 0/47 | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 3/47 | 3/45 | 3/46 | 3/47 | 6/45 | 6/47 | 4/46 | 7/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (Fasted): Treatment A (N=47) | Part 1 (Fasted): Treatment B (N=45) | Part 1 (Fasted): Treatment C (N=46) | Part 1 (Fasted): Treatment D (N=47) | Part 2 (Fed): Treatment A (N=45) | Part 2 (Fed): Treatment B (N=47) | Part 2 (Fed): Treatment C (N=46) | Part 2 (Fed): Treatment D (N=46)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Psychogenic respiratory distress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.